CLINICAL TRIAL: NCT04868500
Title: Managing Asthma Patients With AMAZE™: A Novel Disease Management Platform, A Clinical Pilot Study
Brief Title: Managing Asthma Patients With AMAZE™: A Novel Disease Management Platform
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: Massachusetts General Hospital (Other); Evidera (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: N4280000000
Record Dates: First submitted 2021-03-17; First posted 2021-05-03 (Actual); Results first posted 2023-02-08 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2023-01

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Massachusetts General Hospital (MGH) Participants (Experimental): Participants will use the AMAZE™ application to enter daily asthma symptoms and impact to communicate this information to their healthcare provider, as well as access disease educational materials up to six months.
  Interventions: Device: AMAZE™ Application
- Massachusetts General Hospital (MGH) Clinical Site Staff (Experimental): Clinical site staff will use the AMAZE™ dashboard for six months to identify usability and barriers, benefits, challenges, ease of implementation, and areas for improvement of the AMAZE™ dashboard in a clinical setting.
  Interventions: Device: AMAZE™ Dashboard

INTERVENTIONS:
Device: AMAZE™ Application — Participants will use the AMAZE™ application to enter daily asthma symptoms and impact to communicate this information to their healthcare provider, as well as access disease educational materials up to six months.
  Arms: Massachusetts General Hospital (MGH) Participants
Device: AMAZE™ Dashboard — Clinical site staff will use the AMAZE™ dashboard for six months to identify usability and barriers, benefits, challenges, ease of implementation, and areas for improvement of the AMAZE™ dashboard in a clinical setting.
  Arms: Massachusetts General Hospital (MGH) Clinical Site Staff

SUMMARY:
The primary study objective is to generate evidence as to the feasibility, usability, perceived value, and potential benefits of implementing the AMAZE™ platform into clinical practice.

DETAILED DESCRIPTION:
AstraZeneca has developed the AMAZE™ disease management platform to be used across multiple disease indications to provide a unified experience for the management of participants throughout their participant care journey. AMAZE™ integrates multiple systems, including a patient mobile application where patients can enter daily symptoms and impact to communicate this information to their healthcare provider, as well as access disease educational materials. Implementation of AMAZE™ within clinical practice has not yet been evaluated. The results from this study will be used to inform any changes or modifications that need to be made to the technology platform, its implementation process, and explore impact on clinical outcomes.

ELIGIBILITY:
Inclusion Criteria:

* >18 years of age at the time of enrollment
* Clinically confirmed diagnosis of asthma
* Access to a smartphone with internet access with the following requirements: iOS (Operating System iOS 13 or newer and Devices iPhone 8 or newer) or Android (Operating System 8.0 or newer)
* Able to understand and speak English sufficiently to be able to use the AMAZE™ patient app
* Willingness to participate in a telephone interview and be audio-recorded
* Consenting to participate in the study

Exclusion Criteria:

* Current diagnosis of active chronic obstructive pulmonary disease (COPD) or any pulmonary diagnosis other than asthma
* Has a cognitive impairment, hearing difficulty, acute psychopathology, medical condition, or insufficient knowledge of the English language that, in the opinion of the investigator, would interfere with his or her ability to agree to participate and/or complete the ACT™.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2021-04-27 (Actual); Primary Completion 2021-11-30 (Actual); Study Completion 2021-11-30 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Research Site, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal. All request will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
  Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the deidentified individual patient-level data in an approved sponsored tool . Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home

REFERENCES:
- [Derived] Alladina J, Moschovis PP, Gandhi HN, Carstens D, Bacci ED, Cutts K, Coyne KS, Goldsborough K, Jiang D, O'Brien C, Bernard Kinane T. Observational study of the Amaze asthma disease management platform. Digit Health. 2024 Oct 22;10:20552076241282380. doi: 10.1177/20552076241282380. eCollection 2024 Jan-Dec. PMID 39479373
- See also: Related Info — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=N4280000000&attachmentIdentifier=68577816-6a4e-44ca-9d9d-5cc363bbd99f&fileName=EVA-28838_AMAZE_Redacted_Synopsis_20July2022_Clean_V2-v1.pdf&versionIdentifier=
- See also: Related Info — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=N4280000000&attachmentIdentifier=1bde190a-9f41-4102-af15-b25bdbb9b4d7&fileName=1_clean_Asthma_Sponsor_Protocol_AZPulm_2021Aug10-Redacted.pdf&versionIdentifier=
- See also: Related Info — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=N4280000000&attachmentIdentifier=f209dddf-4104-405b-983f-7c7e39d6d2ef&fileName=EVA-28838_AMAZE_DMP_SAP_v5.0_27July2021_FINAL-Redacted.pdf&versionIdentifier=

RESULTS

PARTICIPANT FLOW:
Groups:
- Massachusetts General Hospital (MGH) Participants: Participants used the AMAZE™ application to enter daily asthma symptoms and impact to communicate this information to their healthcare provider, as well as access disease educational materials up to six months.
- Massachusetts General Hospital (MGH) Clinical Site Staff: Clinical site staff used the AMAZE™ dashboard for six months to identify usability and barriers, benefits, challenges, ease of implementation, and areas for improvement of the AMAZE™ dashboard in a clinical setting.
Period: Overall Study
Arm/Group | Massachusetts General Hospital (MGH) Participants | Massachusetts General Hospital (MGH) Clinical Site Staff
Started | 42 | 7
Not Started (Participants and Clinical Site Staff who terminated early due to clinician's decision and who never opened the Application (App)) | 4 | 1
Completed | 38 | 6
Not Completed | 4 | 1
Not completed — Participants and Clinical Site Staff terminated early | 3 | 1
Not completed — Participants and Clinical Site Staff never opened App | 1 | 0

BASELINE CHARACTERISTICS:
Population: All eligible participants who successfully enrolled in the implementation study were analyzed.
Groups:
- Total: Total of all reporting groups
Arm/Group | Massachusetts General Hospital (MGH) Participants | Massachusetts General Hospital (MGH) Clinical Site Staff | Total
Number analyzed (Participants) | 38 | 6 | 44
Age, Continuous [Mean (Standard Deviation); unit: Years] — Not recorded for MGH Clinical Site Staff. Population: Data only collected for MGH Participants arm for this baseline measure.
  Years
    number analyzed (Participants) | 38 | 0 | 38
    (all) | 24.5 (12.0) |  | 24.5 (12.0)
Sex: Female, Male [Count of Participants; unit: Participants] — Not recorded for MGH Clinical Site Staff. Population: Data only collected for MGH Participants arm for this baseline measure.
  Participants
    number analyzed (Participants) | 38 | 0 | 38
    Female | 26 | 0 | 26
    Male | 12 | 0 | 12
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Not recorded for MGH Clinical Site Staff. Population: Data only collected for MGH Participants arm for this baseline measure.
  Participants
    number analyzed (Participants) | 38 | 0 | 38
    Hispanic or Latino | 7 |  | 7
    Not Hispanic or Latino | 30 |  | 30
    Unknown or Not Reported | 1 |  | 1
Race (NIH/OMB) [Count of Participants; unit: Participants] — Not recorded for MGH Clinical Site Staff. Population: Data only collected for MGH Participants arm for this baseline measure.
  Participants
    number analyzed (Participants) | 38 | 0 | 38
    American Indian or Alaska Native | 0 |  | 0
    Asian | 0 |  | 0
    Native Hawaiian or Other Pacific Islander | 0 |  | 0
    Black or African American | 2 |  | 2
    White | 33 |  | 33
    More than one race | 0 |  | 0
    Unknown or Not Reported | 3 |  | 3

OUTCOME MEASURES:

1. Primary Outcome: Number of Days Participants Accessed the AMAZE™ App (Weeks 1 to 4)
Description: Participant App usage was measured as the number of days the participant engaged (ie., participants accessed 'Home, Daily asthma log, Air quality, My plan, Trends, Appointments, Educational material, Messages, and Notifications') with the App during Weeks 1 to 4.
Time Frame: Weeks 1 to 4
Population: All eligible participants successfully enrolled in the implementation study were analyzed. Here, 'Number of Participants Analyzed' denotes number of participants who accessed the App for the specified time frame and 'Number Analyzed' denotes number of participants analyzed for the specified parameter.
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Massachusetts General Hospital (MGH) Participants
Number analyzed (Participants) | 36
Days
  Home | 16.8 (7.1)
  Daily asthma log | 16.5 (6.8)
  Air quality: number analyzed (Participants) | 11
  Air quality | 2.3 (1.5)
  My plan: number analyzed (Participants) | 30
  My plan | 2.2 (1.5)
  Trends: number analyzed (Participants) | 26
  Trends | 2.8 (3.0)
  Appointments: number analyzed (Participants) | 4
  Appointments | 1.3 (0.5)
  Educational material: number analyzed (Participants) | 3
  Educational material | 1.0 (0.0)
  Messages: number analyzed (Participants) | 26
  Messages | 2.3 (2.4)
  Notifications: number analyzed (Participants) | 35
  Notifications | 1.3 (0.5)

2. Primary Outcome: Number of Days Participants Accessed the AMAZE™ App (Weeks 5 to 8)
Description: Participant App usage was measured as the number of days the participant engaged (ie., participants accessed 'Home, Daily asthma log, Air quality, My plan, Trends, Appointments, Educational material, Messages, and Notifications') with the App during Weeks 5 to 8.
Time Frame: Weeks 5 to 8
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Massachusetts General Hospital (MGH) Participants
Number analyzed (Participants) | 33
Days
  Home | 12.5 (8.6)
  Daily asthma log | 12.1 (8.6)
  Air quality: number analyzed (Participants) | 2
  Air quality | 1.5 (0.7)
  My plan: number analyzed (Participants) | 15
  My plan | 1.6 (0.8)
  Trends: number analyzed (Participants) | 16
  Trends | 1.6 (0.8)
  Appointments: number analyzed (Participants) | 4
  Appointments | 1.3 (0.5)
  Educational material: number analyzed (Participants) | 2
  Educational material | 1.0 (0.0)
  Messages: number analyzed (Participants) | 13
  Messages | 1.8 (1.5)
  Notifications: number analyzed (Participants) | 2
  Notifications | 1.0 (0.0)

3. Primary Outcome: Number of Days Participants Accessed the AMAZE™ App (Weeks 9 to 12)
Description: Participant App usage was measured as the number of days the participant engaged (ie., participants accessed 'Home, Daily asthma log, Air quality, My plan, Trends, Appointments, Educational material, Messages, and Notifications') with the App during Weeks 9 to 12.
Time Frame: Weeks 9 to 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Massachusetts General Hospital (MGH) Participants
Number analyzed (Participants) | 30
Days
  Home | 11.4 (8.1)
  Daily asthma log: number analyzed (Participants) | 29
  Daily asthma log | 11.2 (7.8)
  Air quality: number analyzed (Participants) | 2
  Air quality | 1.0 (0.0)
  My plan: number analyzed (Participants) | 11
  My plan | 1.5 (1.0)
  Trends: number analyzed (Participants) | 9
  Trends | 1.4 (0.5)
  Appointments: number analyzed (Participants) | 3
  Appointments | 1.3 (0.6)
  Educational material: number analyzed (Participants) | 1
  Educational material | 1.0 (NA) — Standard deviation was not reported as only one participant was evaluable for the specified arm group.
  Messages: number analyzed (Participants) | 13
  Messages | 1.4 (0.5)
  Notifications: number analyzed (Participants) | 4
  Notifications | 1.0 (0.0)

4. Primary Outcome: Number of Days Participants Accessed the AMAZE™ App (Weeks 13 to 16)
Description: Participant App usage was measured as the number of days the participant engaged (ie., participants accessed 'Home, Daily asthma log, Air quality, My plan, Trends, Appointments, Educational material, Messages, and Notifications') with the App during Weeks 13 to 16.
Time Frame: Weeks 13 to 16
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Massachusetts General Hospital (MGH) Participants
Number analyzed (Participants) | 25
Days
  Home | 12.6 (8.2)
  Daily asthma log | 12.1 (8.1)
  Air quality: number analyzed (Participants) | 3
  Air quality | 1.0 (0.0)
  My plan: number analyzed (Participants) | 10
  My plan | 1.1 (0.3)
  Trends: number analyzed (Participants) | 12
  Trends | 1.1 (0.3)
  Appointments: number analyzed (Participants) | 5
  Appointments | 1.2 (0.4)
  Educational material: number analyzed (Participants) | 3
  Educational material | 1.0 (0.0)
  Messages: number analyzed (Participants) | 12
  Messages | 1.3 (0.6)
  Notifications: number analyzed (Participants) | 2
  Notifications | 1.0 (0.0)

5. Primary Outcome: Number of Days Participants Accessed the AMAZE™ App (Weeks 17 to 20)
Description: Participant App usage was measured as the number of days the participant engaged (ie., participants accessed 'Home, Daily asthma log, Air quality, My plan, Trends, Appointments, Educational material, Messages, and Notifications') with the App during Weeks 17 to 20.
Time Frame: Weeks 17 to 20
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Massachusetts General Hospital (MGH) Participants
Number analyzed (Participants) | 22
Days
  Home | 9.3 (7.5)
  Daily asthma log | 8.9 (7.2)
  Air quality: number analyzed (Participants) | 1
  Air quality | 1.0 (NA) — Standard deviation was not reported as only one participant was evaluable for the specified arm group.
  My plan: number analyzed (Participants) | 5
  My plan | 1.2 (0.4)
  Trends: number analyzed (Participants) | 6
  Trends | 1.2 (0.4)
  Appointments: number analyzed (Participants) | 2
  Appointments | 1.5 (0.7)
  Educational material: number analyzed (Participants) | 1
  Educational material | 1.0 (NA) — Standard deviation was not reported as only one participant was evaluable for the specified arm group.
  Messages: number analyzed (Participants) | 6
  Messages | 1.3 (0.8)
  Notifications: number analyzed (Participants) | 3
  Notifications | 1.0 (0.0)

6. Primary Outcome: Number of Days Participants Accessed the AMAZE™ App (Weeks 21 to 24)
Description: Participant App usage was measured as the number of days the participant engaged (ie., participants accessed 'Home, Daily asthma log, Air quality, My plan, Trends, Appointments, Educational material, Messages, and Notifications') with the App during Weeks 21 to 24.
Time Frame: Weeks 21 to 24
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Massachusetts General Hospital (MGH) Participants
Number analyzed (Participants) | 14
Days
  Home | 7.6 (7.2)
  Daily asthma log: number analyzed (Participants) | 13
  Daily asthma log | 7.8 (7.3)
  Air quality: number analyzed (Participants) | 0
  My plan: number analyzed (Participants) | 5
  My plan | 1.2 (0.4)
  Trends: number analyzed (Participants) | 3
  Trends | 1.0 (0.0)
  Appointments: number analyzed (Participants) | 1
  Appointments | 3.0 (NA) — Standard deviation was not reported as only one participant was evaluable for the specified arm group.
  Educational material: number analyzed (Participants) | 0
  Messages: number analyzed (Participants) | 4
  Messages | 1.3 (0.5)
  Notifications: number analyzed (Participants) | 0

7. Primary Outcome: Number of Days Clinical Site Staff Accessed the AMAZE™ Dashboard (Weeks 1 to 4)
Description: Clinician dashboard usage was measured as the mean number of days that the clinical site staff accessed the AMAZE™ dashboard during Weeks 1 to 4.
Time Frame: Weeks 1 to 4
Population: Clinical site staff who used the AMAZE™ dashboard at the specified time frame were considered for this outcome measure.
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Massachusetts General Hospital (MGH) Clinical Site Staff
Number analyzed (Participants) | 3
Days | 8.3 (6.7)

8. Primary Outcome: Number of Days Clinical Site Staff Accessed the AMAZE™ Dashboard (Weeks 5 to 8)
Description: Clinician dashboard usage was measured as the mean number of days that the clinical site staff accessed the AMAZE™ dashboard during Weeks 5 to 8.
Time Frame: Weeks 5 to 8
Population: Clinical site staff who used the AMAZE™ dashboard at the specified time frame were considered for this outcome measure.
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Massachusetts General Hospital (MGH) Clinical Site Staff
Number analyzed (Participants) | 5
Days | 5.8 (6.1)

9. Primary Outcome: Number of Days Clinical Site Staff Accessed the AMAZE™ Dashboard (Weeks 9 to 12)
Description: Clinician dashboard usage was measured as the mean number of days that the clinical site staff accessed the AMAZE™ dashboard during Weeks 9 to 12.
Time Frame: Weeks 9 to 12
Population: Clinical site staff who used the AMAZE™ dashboard at the specified time frame were considered for this outcome measure.
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Massachusetts General Hospital (MGH) Clinical Site Staff
Number analyzed (Participants) | 5
Days | 6.6 (6.1)

10. Primary Outcome: Number of Days Clinical Site Staff Accessed the AMAZE™ Dashboard (Weeks 13 to 16)
Description: Clinician dashboard usage was measured as the mean number of days that the clinical site staff accessed the AMAZE™ dashboard during Weeks 13 to 16.
Time Frame: Weeks 13 to 16
Population: Clinical site staff who used the AMAZE™ dashboard at the specified time frame were considered for this outcome measure.
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Massachusetts General Hospital (MGH) Clinical Site Staff
Number analyzed (Participants) | 6
Days | 5.8 (6.5)

11. Primary Outcome: Number of Days Clinical Site Staff Accessed the AMAZE™ Dashboard (Weeks 17 to 20)
Description: Clinician dashboard usage was measured as the mean number of days that the clinical site staff accessed the AMAZE™ dashboard during Weeks 17 to 20.
Time Frame: Weeks 17 to 20
Population: Clinical site staff who used the AMAZE™ dashboard at the specified time frame were considered for this outcome measure.
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Massachusetts General Hospital (MGH) Clinical Site Staff
Number analyzed (Participants) | 5
Days | 5.6 (6.5)

12. Primary Outcome: Number of Days Clinical Site Staff Accessed the AMAZE™ Dashboard (Weeks 21 to 24)
Description: Clinician dashboard usage was measured as the mean number of days that the clinical site staff accessed the AMAZE™ dashboard during Weeks 21 to 24.
Time Frame: Weeks 21 to 24
Population: Clinical site staff who used the AMAZE™ dashboard at the specified time frame were considered for this outcome measure.
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Massachusetts General Hospital (MGH) Clinical Site Staff
Number analyzed (Participants) | 3
Days | 6.7 (4.9)

13. Primary Outcome: Number of Participants Engaged in Agreement of Visit Survey Item 9 (Weeks 1 to 4)
Description: Visit Survey Item 9 was 'The visit helped avoid an emergency room (ER) or urgent care center visit or hospitalization.' Visit surveys were completed throughout the study whenever a participant completed an asthma-related clinic visit. Number of participants engaged in agreement of Visit Survey Item 9 as 'High' (ie., 5-7 days per week per month) and 'Very low' (ie., less than one day per week per month) are reported.
Time Frame: Weeks 1 to 4
Population: All eligible participants successfully enrolled in the implementation study were analyzed. Here, 'Number of Participants Analyzed' denotes number of participants analyzed for the specified time frame.
Measure: Count of Participants; unit: Participants
Arm/Group | Massachusetts General Hospital (MGH) Participants
Number analyzed (Participants) | 1
Participants
  High | 1
  Very low | 0

14. Primary Outcome: Number of Participants Engaged in Agreement of Visit Survey Item 9 (Weeks 5 to 8)
Description: Visit Survey Item 9 was 'The visit helped avoid an ER or urgent care center visit or hospitalization.' Visit surveys were completed throughout the study whenever a participant completed an asthma-related clinic visit. Number of participants engaged in agreement of Visit Survey Item 9 as 'High' (ie., 5-7 days per week per month) and 'Very low' (ie., less than one day per week per month) are reported.
Time Frame: Weeks 5 to 8
Population: as for outcome 13
Measure: Count of Participants; unit: Participants
Arm/Group | Massachusetts General Hospital (MGH) Participants
Number analyzed (Participants) | 1
Participants
  High | 1
  Very low | 0

15. Primary Outcome: Number of Participants Engaged in Agreement of Visit Survey Item 9 (Weeks 9 to 12)
Description: as for outcome 14
Time Frame: Weeks 9 to 12
Population: as for outcome 13
Measure: Count of Participants; unit: Participants
Arm/Group | Massachusetts General Hospital (MGH) Participants
Number analyzed (Participants) | 1
Participants
  High | 1
  Very low | 0

16. Primary Outcome: Number of Participants Engaged in Agreement of Visit Survey Item 9 (Weeks 13 to 16)
Description: as for outcome 14
Time Frame: Weeks 13 to 16
Population: as for outcome 13
Measure: Count of Participants; unit: Participants
Arm/Group | Massachusetts General Hospital (MGH) Participants
Number analyzed (Participants) | 1
Participants
  High | 1
  Very low | 0

17. Primary Outcome: Number of Participants Engaged in Agreement of Visit Survey Item 9 (Weeks 17 to 20)
Description: as for outcome 14
Time Frame: Weeks 17 to 20
Population: as for outcome 13
Measure: Count of Participants; unit: Participants
Arm/Group | Massachusetts General Hospital (MGH) Participants
Number analyzed (Participants) | 1
Participants
  High | 0
  Very low | 1

18. Primary Outcome: Number of Participants Engaged in Agreement of Visit Survey Item 9 (Weeks 21 to 24)
Description: as for outcome 14
Time Frame: Weeks 21 to 24
Population: No participant completed at least one daily asthma log during the specified time frame (Weeks 21 to 24), so no data was reported.
Arm/Group | Massachusetts General Hospital (MGH) Participants
Number analyzed (Participants) | 0

19. Primary Outcome: Evaluate Participant Satisfaction With the AMAZE™ App (End of Study)
Description: Satisfaction with the AMAZE™ App features was measured by the number of participants who reported satisfaction on parameters of 'Very unsatisfied, Unsatisfied, Neutral, Satisfied, and Very satisfied'.
Time Frame: End of Study (Month 6)
Population: All eligible participants successfully enrolled in the implementation study were analyzed. Here, 'Number of Participants Analyzed' denotes number of participants analyzed at Month 6.
Measure: Count of Participants; unit: Participants
Arm/Group | Massachusetts General Hospital (MGH) Participants
Number analyzed (Participants) | 22
Participants
  Very unsatisfied | 1
  Unsatisfied | 0
  Neutral | 3
  Satisfied | 12
  Very satisfied | 6

20. Primary Outcome: Emergency Room Visits, Urgent Care Center Visits, or Hospitalization Avoidance (End of Study)
Description: The impact of AMAZE™ on ER, urgent care center visits, and hospitalizations was measured as the number of participants who reported "agree" or "strongly agree" with the question 'Since the start of the study, use of the AMAZE™ App helped me avoid ER or urgent care center visits or hospitalizations.' from the participant visit experience survey.
Time Frame: End of Study (Month 6)
Population: as for outcome 19
Measure: Count of Participants; unit: Participants
Arm/Group | Massachusetts General Hospital (MGH) Participants
Number analyzed (Participants) | 22
Participants
  Strongly agree | 2
  Agree | 1

21. Primary Outcome: Impact of AMAZE™ App on Participants Clinic Visits
Description: Visit Survey Item 9 was 'The visit helped avoid an ER or urgent care center visit or hospitalization.' The impact of AMAZE™ on participant visits was measured as the number of participants who selected "agree" or "strongly agree" in response to the 9-items in the participant visit experience survey.
Time Frame: Day 1 through End of Study (Month 6)
Population: as for outcome 13
Measure: Count of Participants; unit: Participants
Arm/Group | Massachusetts General Hospital (MGH) Participants
Number analyzed (Participants) | 20
Participants
  Strongly agree | 2
  Agree | 0

22. Primary Outcome: Participant Perception of Appointment Discussions and Taking Part in Asthma Decisions (End of Study)
Description: The impact of AMAZE™ on improved participant communication with their healthcare provider was measured as the number of participants who reported "agree" or "strongly agree" with the questions "The app helped me discuss my asthma with my healthcare providers during my most recent visit?", "App helped the appointment with my doctor go more smoothly?" and "I was included in making decisions about my asthma treatment during my most recent visit?" on the participant visit experience survey.
Time Frame: End of Study (Month 6)
Population: as for outcome 19
Measure: Count of Participants; unit: Participants
Arm/Group | Massachusetts General Hospital (MGH) Participants
Number analyzed (Participants) | 20
Participants
  Asthma discussions-Strongly Agree | 3
  Asthma Discussions-Agree | 5
  To take appointment smoothly-Strongly agree | 3
  To take appointment smoothly-Agree | 3
  Asthma treatment decision-Strongly agree | 14
  Asthma treatment decision-Agree | 4

23. Primary Outcome: Patient Satisfaction Questionnaire-18 Subscale Scores (End of Study)
Description: Participant satisfaction with their healthcare experience was evaluated using the PSQ-18 items with subscale scores of 'General satisfaction, Technical quality, Interpersonal manner, Communication, Financial aspects, Time spent with doctor, Accessibility and convenience' at End of Study (Month 6). The PSQ-18 scores ranges from 1 to 5 and a higher score indicates greater satisfaction.
Time Frame: End of study (Month 6)
Population: as for outcome 19
Measure: Mean (Standard Deviation); unit: Scores on a Scale
Arm/Group | Massachusetts General Hospital (MGH) Participants
Number analyzed (Participants) | 22
Scores on a Scale
  General satisfaction | 4.1 (0.86)
  Technical quality | 4.3 (0.61)
  Interpersonal manner | 4.3 (0.57)
  Communication | 4.2 (0.77)
  Financial aspects | 4.0 (0.91)
  Time spent with doctor | 3.8 (0.95)
  Accessibility and convenience | 3.6 (0.89)

24. Primary Outcome: Patient-Reported System Usability Scale (SUS) (Month 1)
Description: The usability of the AMAZE™ App was measured by the number of participants who rated the app as 'excellent, good, okay, poor, awful or skipped to report' at Month 1.
Time Frame: Month 1
Population: All eligible participants successfully enrolled in the implementation study were analyzed. Here, 'Number of Participants Analyzed' denotes number of participants analyzed at Month 1.
Measure: Count of Participants; unit: Participants
Arm/Group | Massachusetts General Hospital (MGH) Participants
Number analyzed (Participants) | 30
Participants
  Excellent | 17 (56.7)
  Good | 9 (30.0)
  Okay | 0 (0.0)
  Poor | 3 (10.0)
  Awful | 0 (0.0)
  Skipped | 1 (3.3)

25. Primary Outcome: Patient-Reported SUS (End of Study)
Description: The usability of the AMAZE™ App was measured by the number of participants who rated the app as 'excellent, good, okay, poor, awful or skipped to report' at End of Study (Month 6).
Time Frame: End of Study (Month 6)
Population: as for outcome 19
Measure: Count of Participants; unit: Participants
Arm/Group | Massachusetts General Hospital (MGH) Participants
Number analyzed (Participants) | 22
Participants
  Excellent | 14 (63.6)
  Good | 6 (27.3)
  Okay | 0 (0.0)
  Poor | 0 (0.0)
  Awful | 2 (9.1)
  Skipped | 0 (0.0)

26. Primary Outcome: Clinical Site Staff-Reported SUS (Month 1)
Description: The usability of the AMAZE™ dashboard was measured by the number of clinical staff who rated the App as 'excellent, good, okay, poor, awful or skipped to report' at Month 1.
Time Frame: Month 1
Population: Clinical site staff who used the AMAZE™ dashboard at the specified time frame were considered for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Massachusetts General Hospital (MGH) Clinical Site Staff
Number analyzed (Participants) | 5
Participants
  Excellent | 0 (0.0)
  Good | 4 (80.0)
  Okay | 0 (0.0)
  Poor | 1 (20.0)
  Awful | 0 (0.0)
  Skipped | 0 (0.0)

27. Primary Outcome: Clinical Site Staff-Reported SUS (End of Study)
Description: The usability of the AMAZE™ dashboard was measured by the number of clinical staff who rated the App as 'excellent, good, okay, poor, awful or skipped to report' at End of Study (Month 6).
Time Frame: End of Study (Month 6)
Population: Clinical site staff who used the AMAZE™ dashboard at the specified time frame were considered for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Massachusetts General Hospital (MGH) Clinical Site Staff
Number analyzed (Participants) | 4
Participants
  Excellent | 1 (25.0)
  Good | 1 (25.0)
  Okay | 0 (0.0)
  Poor | 1 (25.0)
  Awful | 0 (0.0)
  Skipped | 1 (25.0)

28. Primary Outcome: Evaluate Ease of Implementation of AMAZE™ App in Clinical Setting (End of Study)
Description: The ease of implementation of AMAZE™ was measured by the number of clinical staff who reported "very easy" or "somewhat easy" to the question "How would you rate the overall ease of implementing AMAZE™ on a platform into your clinical practice?" in the post-study survey at End of Study (Month 6).
Time Frame: End of Study (Month 6)
Population: Clinical site staff who used the AMAZE™ dashboard at the specified time frame were considered for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Massachusetts General Hospital (MGH) Clinical Site Staff
Number analyzed (Participants) | 6
Participants
  Very easy | 4
  Somewhat easy | 0

29. Primary Outcome: Evaluate Impact of AMAZE™ App on Managing Participants (End of Study)
Description: The impact of AMAZE™ on managing participants was measured by the number of clinical staff who reported "moderately" or "very well" to the question "Did the AMAZE™ help you manage your participants?" in the post-study survey at End of Study (Month 6).
Time Frame: End of Study (Month 6)
Population: Clinical site staff who used the AMAZE™ dashboard at the specified time frame were considered for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Massachusetts General Hospital (MGH) Clinical Site Staff
Number analyzed (Participants) | 6
Participants
  Moderately | 2
  Very well | 0

30. Primary Outcome: Evaluate Perceived Benefit of AMAZE™ App in Clinical Setting (End of Study)
Description: The perceived benefit of AMAZE™ was evaluated by the number of clinical staff who endorsed different perceived benefits as "Ability to track symptoms, Ability to track asthma triggers, Ability to track reliever medication use, Ability track ER visits/ hospitalizations, and Integration of AMAZE™ platform with electronic health records" based on the item "What did you find the most useful about the AMAZE™ platform?" in the post-study survey at End of Study (Month 6).
Time Frame: End of Study (Month 6)
Population: Clinical site staff who used the AMAZE™ dashboard at the specified time frame were considered for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Massachusetts General Hospital (MGH) Clinical Site Staff
Number analyzed (Participants) | 6
Participants
  Ability to track symptoms | 2
  Ability to track asthma triggers | 1
  Ability to track reliever medication use | 2
  Ability track ER visits/ hospitalizations | 0
  Integration of AMAZE™ platform with electronic health records | 2

31. Primary Outcome: Evaluate Perceived Disadvantages of AMAZE™ in Clinical Setting (End of Study)
Description: The perceived disadvantages of AMAZE™ were evaluated by the number of clinical site staff who endorsed different perceived disadvantages as "Ability to track air flow measurements, Participant-health care provides (HCP) messaging feature, Ability to assign another healthcare provider to a participant, Ability to track level of impairment through Asthma Control Test (ACT™) scores" based on the question "What did you find the least useful or cumbersome about the AMAZE™ platform?" in the post-study survey at End of Study (Month 6).
Time Frame: End of Study (Month 6).
Population: Clinical site staff who used the AMAZE™ dashboard at the specified time frame were considered for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Massachusetts General Hospital (MGH) Clinical Site Staff
Number analyzed (Participants) | 6
Participants
  Ability to track air flow measurements | 1
  Participant-HCP messaging feature | 2
  Ability to assign another healthcare provider to a participant | 1
  Ability to track level of impairment through ACT™ scores | 1

ADVERSE EVENTS:
Time Frame: All-Cause Mortality, Serious, and Other (Not Including Serious) Adverse Events were not monitored/assessed.
Description: This was an interventional study with no requirements to collect adverse events during the study since enrollment in the study was based on disease diagnosis and did not require the administration of a study drug. All-Cause Mortality, Serious, and Other (Not Including Serious) Adverse Events were not monitored/assessed.
Arm/Group | Massachusetts General Hospital (MGH) Participants | Massachusetts General Hospital (MGH) Clinical Site Staff
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
This was an interventional study with no requirements to collect adverse events during the study since enrollment in the study was based on disease diagnosis and did not require the administration of a study drug.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
MedImmune has 60 days to review results communications prior to public release and may delete information that compromises ongoing studies or is considered proprietary. This restriction is not intended to compromise the objective scientific integrity of the manuscript, it being understood that results shall be published regardless of outcome.

DOCUMENTS (2):
  • Study Protocol (2021-08-10): https://cdn.clinicaltrials.gov/large-docs/00/NCT04868500/Prot_000.pdf
  • Statistical Analysis Plan (2021-07-27): https://cdn.clinicaltrials.gov/large-docs/00/NCT04868500/SAP_001.pdf